CLINICAL TRIAL: NCT01689610
Title: Non-Interventional Study to Investigate Efficacy and Safety of Nab-Paclitaxel in Patients With Metastatic Breast Cancer
Brief Title: Non-interventional Study With Nab-Paclitaxel (Abraxane®)
Acronym: NABUCCO
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-02240
Record Dates: First submitted 2012-08-14; First posted 2012-09-21 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Metastatic Breast Cancer
Keywords: Nab-Paclitaxel; Abraxane; Nabucco; safety; breast cancer; daily routine; peripheral neuropathy; iOMEDICO
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult female patients with MBC: This is an observational study, no interventions are specified

SUMMARY:
The purpose of this non-interventional study is to collect data on the efficacy and safety of Nab-Paclitaxel in the routine application.

DETAILED DESCRIPTION:
The main focus of this non-interventional study is set on answering the following questions:

* Can the results observed in controlled clinical trials regarding efficacy and safety be reproduced in the routine clinical setting?
* Are the side-effects of nab-paclitaxel therapy observed in this study comparable to the previously described safety-profile in terms of frequency and intensity?
* What are the main reasons for modification or termination of the nab-paclitaxel therapy?
* How does nab-paclitaxel therapy influence the patients' quality of life?
* What are the criteria for selecting nab-paclitaxel as therapy for metastatic breast cancer?

ELIGIBILITY:
Inclusion Criteria:

* Female Patients with metastatic breast cancer, who are at least 18 years old (no upper age limit)

Exclusion Criteria:

* Contraindication according to the summary of product characteristics of Abraxane®
* No signed patient informed consent form available
* pregnant or breastfeeding patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients with metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 705 (Actual)
Dates: Start 2012-04; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Time to Tumor Progression (TTP) | 6 months after last-patient-in (LPI)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 6 months after last-patient-in (LPI)
Overall survival (OS) | 6 months after last-patient-in (LPI)
Time to treatment discontinuation | 6 months after last-patient-in (LPI)
Number of participants with Adverse Events as a measure of safety and tolerability | Until 30 days after discontinuation of Nab-paclitaxel
Relative dosage of Nab-Paclitaxel | Until discontinuation of Nab-Paclitaxel, up to 6 month
Intensity of peripheral neuropathy | Until discontinuation of Nab-Paclitaxel, up to 6 month
Occurence of neutropenia | Until discontinuation of Nab-Paclitaxel, up to 6 month
Necessity of supportive medication (e.g. haematopoetic growth factors, analgetics, antibiotics and antiemetics) | Until discontinuation of Nab-Paclitaxel, up to 6 month
Patient reported outcome on Quality of life and adverse events | At baseline, 3 and 6 months after start of treatment
  Assessed by questionnaires FACT-G, FACT-B, FACT-Taxanes and a pain questionnaire of the Robert-Koch-Institute.
Reasons for dose modifications or discontinuation of treatment | Until discontinuation of Nab-Paclitaxel, up to 6 month
Occurence of febrile neutropenia | Until discontinuation of Nab-Paclitaxel, up to 6 month
Occurence of peripheral neuropathy | Until discontinuation of Nab-Paclitaxel, up to 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Salat, Prof., Principal Investigator — Haemato-Onkologische Schwerpunktpraxis Franz-Schrank-Strasse 2 80638 Munich, Germany
Locations (1):
- iOMEDICO AG, Freiburg im Breisgau, Baden-Wurttemberg, Germany